CLINICAL TRIAL: NCT01320995
Title: Perineal Echography in the Delivery Room for the Detection of Anal Lesions Among Primiparous Mothers: a Randomized Study
Brief Title: Perineal Echography in the Delivery Room for the Detection of Anal Lesions
Acronym: OASIS 1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI/2010/VL-02; 2011-A00050-41 (Other: RCB number)
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Parturition
Keywords: Second degree vaginal tear; Perineal ultrasound; Anal incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental arm (Experimental): In this arm, perineal ultrasound is used directly after delivery in order to hypothetically better detect anal lesions.
  Interventions: Procedure: Perineal ultrasound
- Standard arm (No Intervention): No perineal ultrasound immediately after delivery.

INTERVENTIONS:
Procedure: Perineal ultrasound — Perineal ultrasound is performed after delivery in order to better detect sphincter lesions.
  Arms: Experimental arm

SUMMARY:
The main objective of this study is to compare the rate of anal incontinence (measured by the Wexner score, qualitative and quantitative (> 4)) at 3 months post partum among primiparas with vaginal tears ≥ 2nd degree who receive a sphincter injury screening at delivery by conducting a sphincter ultrasound in the delivery room versus a similar group of women who do not benefit from screening.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow up
* The patient is delivering her first child; vaginal delivery
* The patient has a minimum stage 2 perineal lesion
* The patient accepts perineal echography

Exclusion Criteria:

* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Cesarien section
* No perineal lesion (intact perineum)
* Emergency situation which hinders screening for anal lesions under good medical conditions
* Previous vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Presence/absence of anal incontinence | 3 months
  Anal incontinence is defined as a Wexner score > 4

SECONDARY OUTCOMES:
Wexner anal incontinence score | 3 months
Visual Analog Scale for discomfort during perineal ultrasound | 2 hours
  Ranges from 0.0 to 10.0
Kappa coefficient for second reading of ultrasounds | 30 days
  A second reading of each ultrasound is obtained within 30 days. The Kappa coefficient of concordance will be calculated between the two readings.
Presence/absence of a sphincter tear | 2 hours
  Presence/absence of a sphincter tear immediately after delivery.
Patient requires anal sutures (yes/no) | 2 hours
  Patient requires anal sutures after delivery?
Presence/absence of suture infection | 3 months
  Has an infection ocurred between delivery and the follow up visit at 3 months post partum?
Questionnaire PFIQ | 3 months
Questionnaire PFDI | 3 months
Questionnaire SF36 | 3 months
Questionnaire Euroqol | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - CHU de Montpellier, Montpellier